CLINICAL TRIAL: NCT02169505
Title: Safety and Efficacy of Brentuximab Vedotin Maintenance After Allogeneic and Haploidentical Stem Cell Transplantation in High Risk CD30+ Lymphoma (Hodgkin Lymphoma and ALCL)
Brief Title: Brentuximab Vedotin in High-Risk CD30+ Lymphoma Post Allogeneic Stem Cell Transplantation (AlloSCT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0351; NCI-2014-01593 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-06-11; First posted 2014-06-23 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma
Keywords: Lymphoma; Hodgkin lymphoma; HL; CD30 positive Hodgkin Lymphoma; Anaplastic large cell lymphoma; ALCL; Allogeneic Stem Cell Transplantation; ASCT; Graft-versus-host disease; GVHD; Brentuximab Vedotin; SGN-35; Adcetris
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Graft vs Host Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin (Experimental): Brentuximab by vein over 30 minutes every 3 weeks for a total of 6 cycles starting between days 30 and 60 post allogeneic stem cell transplant (SCT).
  Brentuximab dose based on actual body weight starting with an initial dose of 1.2 mg/kg for the first 2 cycles and dose increased to 1.8 mg/kg after the second cycle for all subsequent cycles.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Starting dose: 1.2 mg/kg by vein on Day 1 for the first 2, 21 day cycles. Dose increased to 1.8 mg/kg by vein after the second cycle for all subsequent cycles.
  Other Names: SGN-35; Adcetris

SUMMARY:
The goal of this clinical research study is to study the safety of ADCETRISTM (brentuximab vedotin) in patients with Hodgkin lymphoma or ALCL who have had an allogeneic or haploidentical stem cell transplant. Another goal of this study is to learn if brentuximab vedotin can help to prevent the disease from coming back.

DETAILED DESCRIPTION:
Study Drug Administration:

If you agree to take part in this study, about 35-60 days after the transplant, you will receive brentuximab vedotin by vein over about 30 minutes on Day 1 of each 21-day study cycle. You may receive up to 6 cycles of brentuximab vedotin.

At Cycles 3 and beyond, you will receive a higher dose of the study drug than you received during Cycles 1 and 2.

Study Visits:

About 5 days before Day 1 of Cycle 1:

* You will have a physical exam. As part of the physical exam, you will be checked for graft-versus-host disease (GVHD -- when transplanted donor tissue attacks the tissues of the recipient's body). You may have an additional blood draw to check for GVHD as part of your standard of care.
* Blood (about 2 tablespoons) will be drawn for routine tests and to check how the transplant has taken.
* Blood (about 2 teaspoons each time) will be drawn before and after your dose of study drug to check the immune system.

On Days 3 and 5 of Cycle 1, blood (about 2 teaspoons) will be drawn to check the immune system.

About 5 days before Day 1 of Cycles 2-6:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests and to check the immune system.

If your doctor thinks it is needed, you may have a skin biopsy or endoscopy to check for GVHD and/or graft failure. You will sign a separate consent form that explains the procedures and risks.

Length of Study:

You will be taken off study 1 year after the transplant. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, if you develop an infection (such as cytomegalovirus [CMV] that does not respond to treatment), or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Follow-Up Visits:

About 1, 3, 6, and 12 months after the transplant, you will have follow-up visits as part of your standard of care after your transplant. At these visits:

* You will have a physical exam
* Blood (about 4 tablespoons) will be drawn for routine tests, to learn how the transplant has taken, and to check the status of the disease.
* You will have a computed tomography (CT) scan to check the status of the disease.
* You will have a bone marrow biopsy and aspiration to check the status of the disease and for cytogenetic testing. To collect a bone marrow biopsy/aspirate, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. Cytogenetic testing looks at how genetic changes to cells may affect how the disease may react to the study drug.

This is an investigational study. Brentuximab vedotin is FDA approved and commercially available for the treatment of Hodgkin lymphoma and ALCL. It is investigational to give brentuximab vedotin at an earlier time after a transplant.

Up to 20 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD30 positive Hodgkin Lymphoma (HL) or anaplastic large cell lymphoma (ALCL) that have undergone allogeneic or haploidentical SCT in the past 60 days (matched related or matched unrelated donors only).
2. Age 18 to 65 years.
3. Performance status: Zubrod 0-1 or Karnofsky 80-100.
4. Serum creatinine < 1.5 mg/dL or creatinine clearance greater than or equal to 40 cc/min as defined by MDRD method from National Kidney Disease Education Program (NKDEP).
5. Serum direct bilirubin < 1.5 mg/dL (unless Gilbert's syndrome).
6. SGPT < 200 IU/L unless related to patient's malignancy.
7. Evidence of neutrophil and platelet engraftment, defined as platelet count equal or greater than 50,000 mm3 independent of platelet transfusion and ANC equal or greater to 1000 without growth factor support for at least 5 days.
8. Patients with previous exposure to brentuximab pre-transplant are eligible for the study.

Exclusion Criteria:

1. Pregnancy or breast-feeding (women of childbearing potential, any female who has experienced menarche and who has not undergone surgical sterilization or is post-menopausal with a positive serum pregnancy test.
2. Presence of steroid-refractory acute graft-versus-host disease (GVHD).
3. Patients that underwent allogeneic transplantation as a treatment of graft failure.
4. Dual refractory CMV reactivation to foscarnet and ganciclovir or evidence of CMV disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sairah Ahmed, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who have had an Allogeneic and Haploidentical Stem Cell Transplantation in High Risk CD30+ Lymphoma (Hodgkin Lymphoma and ALCL)
Groups:
- Safety and Efficacy of Brentuximab Vedotin Maintenance After A: Study the safety of Brentuximab in patients with HL or ALCL who have had an allo or haplo stem cell transplant. Also learn if drug prevents the disease from coming back.
Period: Overall Study
Arm/Group | Safety and Efficacy of Brentuximab Vedotin Maintenance After A
Started | 2
Completed | 1
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Safety and Efficacy of Brentuximab Vedotin Maintenance After A
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Secondary Graft Failure
Description: Safety is defined by no more than two secondary graft failures within 6 months of transplant (Day 0), based on an observed graft failure rate of <10% using standard of care treatment. If at any time more than two of these events are observed during the specified time frame, the study will be stopped and no further patients will be accrued.
Time Frame: An average of 12 months
Measure: Number; unit: participants
Groups:
- 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6: Dose will be reduced from 1.8 mg/kg to 1.2 mg/kg or from 1.2 mg/kg to 1 mg/kg or from 1 mg/kg to stop treatment if:
  1. Neutropenia grade 3-4 unresponsive to G-CSF or grade 4 thrombocytopenia are observed.
  2. Peripheral neuropathy, new or worsening grade 2 or 3. Withhold treatment until improvement or return to grade 1 or baseline; then resume with a dose reduction.
  Dose will be reduced to 1 mg/kg if:
  1. Creatinine clearance < 30 cc/min as defined by MDRD method from NKDEP. http://nkdep.nih.gov/lab-evaluation/gfr/estimating.shtml
  2. Hepatic impairment defined as bilirubin > 2 mg/dL.
  If the patient develops grade 3-4 neutropenia unresponsive to G-CSF: Hold until resolution to grade </= 1 and restart at lower dose.
Arm/Group | 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6
Number analyzed (Participants) | 1
participants | 0

2. Secondary Outcome: Number of Participants With Hematologic Toxicity
Description: The most common grade > 3 side effects on Brentuximab.
Time Frame: an average of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Number of Participants With Relapse
Description: Evaluate the safety of brentuximab early after allogeneic stem cell transplant and haploidentical allogeneic transplantant and observe if there is a decrease in the risk of relapse.
Time Frame: an average of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Number of Participants With Incidence of Cytomegalovirus (CMV) Reactivation and/or CMV Disease.
Description: Evaluate the CMV in blood
Time Frame: an average of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6
Number analyzed (Participants) | 1
Participants | 0

5. Secondary Outcome: Number of Participants With Acute Graft-versus-host Disease (GVHD).
Description: The tissue and serum in participants were measured by the GVHD
Time Frame: an average of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Number of Participants With Central and Effector Cell Effects
Description: We will perform on peripheral blood for mononuclear cells (PBMC) and serum collected from participants at baseline (prior to initiation of brentuximab therapy) and on days 1, 3, and 5 after initiation of brentuximab and every 21 days thereafter to assess the effect on T cell subsets and their effector function as well as other immune subsets.
Time Frame: an average of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6
Number analyzed (Participants) | 1
Participants | 0

7. Secondary Outcome: Number of Participants With Change in Serum CD30 Levels After Brentuximab Administration
Description: Immunological correlative studies on peripheral blood mononuclear cells (PBMC) and serum will be collected from participants at baseline (prior to initiation of brentuximab therapy) and on days 1, 3, and 5 after initiation of brentuximab and every 21 days thereafter to assess the effect on T cell subsets and their effector function as well as CD30 levels.
Time Frame: an average of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6
Number analyzed (Participants) | 1
Participants | 0

8. Secondary Outcome: Number of Participants With Progression-Free Survival and Overall Survival on Brentuximab Maintenance
Description: The Kaplan-Meier (1958) survival curves were used to estimate the overall survival and progression-free survival. Cox proportional hazards regression analysis was used to model the association between overall survival and progression-free survival and disease and demographic covariates of interest.
Time Frame: an average of 12 months
Population: Participant one had a progression free survival and overall survival.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/kg for C1-2 Then 1.8mg/kg for C3-6
Number analyzed (Participants) | 1
Participants
  Overall | 1
  Progression-free survival | 1

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Treatment Arm: 1.2 mg/kg for C1-2 then 1.8mg/kg for C3-6
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=2)
Decreased ANC (Blood and lymphatic system disorders) | 2
Dcreased WBC (Blood and lymphatic system disorders) | 1
Decreased PLT (Blood and lymphatic system disorders) | 1
Skin Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT02169505/Prot_SAP_000.pdf